CLINICAL TRIAL: NCT02040974
Title: Long Term Follow up in Patients Using Immunotherapy: Efficacy and Impact on Quality of Life
Brief Title: Allergen Immunotherapy in Allergic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Demirturk, expert in allergy and immunology, Istanbul University
Other Study IDs: 1978
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinitis
Keywords: immunotherapy, house dust mites, pollens, allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Our aim was to evaluate the effectiveness of subcutaneous allergen immunotherapy with the symptom scores (RSS), visual analog scale (VAS) and medication scores (MS) and the impact on quality of life with rhinoconjunctivitis quality of life questionnaire (RQLQ) in allergic rhinitis patients sensitized to different allergens. Also the development of new sensitizations and asthma during the immunotherapy were determined.

DETAILED DESCRIPTION:
Allergic rhinitis patients sensitized to at least one common aero-allergen who completed a three or five year period of allergen immunotherapy in our outpatient clinic between 2002-2013 were enrolled in the study and patients with allergic rhinitis who received only medical treatment were chosen as the control group. Patients were separated in two groups according to sensitization patterns including pollens or house dust mites. All patients were evaluated before immunotherapy, in the first and the fifth years of treatment and two years after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinitis/asthma

Exclusion Criteria:

* pregnancy,
* malignity,
* autoimmunity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allergic rhinitis patients sensitized to at least one common aero-allergen who completed a three or five year period of allergen immunotherapy in our outpatient clinic between 2002-2013 were enrolled in the study and patients with allergic rhinitis who received only medical treatment were chosen as the control group. Patients were separated in two groups according to sensitization patterns including pollens or house dust mites. All patients were evaluated before immunotherapy, in the first and the fifth years of treatment and two years after the treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2007-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
The improvent of quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Demirturk, Principal Investigator — Istanbul Faculty of Medicine
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)